CLINICAL TRIAL: NCT03196310
Title: Randomized Single Blinded First CMC Osteoarthritis Treatment: Therapy and Bracing Alone vs. Intra-Articular Corticosteroid Injection vs Intra-Articular Leukocyte Depleted Platelet Rich Plasma
Brief Title: Single Blinded First CMC Osteoarthritis Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kettering Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-008
Record Dates: First submitted 2017-06-21; First posted 2017-06-22 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Osteoarthritis Thumb
MeSH Terms: interventions — Adrenal Cortex Hormones; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be blinded to therapy they receive
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- PRP (Experimental): Intra-articular injection of platelet rich plasma.
  Interventions: Drug: Platelet Concentrate
- Corticosteroid (Active Comparator): Intra-articular injection of kenalog.
  Interventions: Drug: Corticosteroid injection
- Normal Saline (Placebo Comparator): Intra-articular injection of normal saline
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Platelet Concentrate — Platelet Rich plasma
  Arms: PRP
Drug: Corticosteroid injection — Kenalog
  Arms: Corticosteroid
Other: Normal Saline — Control Group - Placebo
  Arms: Normal Saline

SUMMARY:
Single blinded PRP vs. Corticosteroid vs. Placebo (normal saline) intra-articular injection for basal joint arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1-3 osteoarthritis of the basal joint

Exclusion Criteria:

* Patients with Stage 4 1st carpometacarpal joint arthritis as described by Eaton
* Patients who have received a corticosteroid injection in the last year to the 1st CMC joint on the proposed study side
* Patients who have scaphotriquetral, radioscaphoid, or scaphotrapezial osteoarthritis
* Patients who have concurrent DeQuervain's tenosynovitis or intersection syndrome or have been treated for either of these in the last 3 months
* Patients undergoing evaluation of cervical radiculopathy
* Patients with fibromyalgia or inflammatory rheumatic disease
* Patients with Pressier disease, Kienbock's, or avascular necrosis of the scaphoid
* Patients with any history of primary or secondary bone tumor
* Patients that are pregnant or terminally ill

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Disabilities arm shoulder and hand score | 1 year
  functional score

SECONDARY OUTCOMES:
Pinch Strength | 1 year
  Objective measurement

OTHER OUTCOMES:
Visual Analog Score | 1 year
  Pain reduction

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopedic Associates of Southwest Ohio, Centerville, Ohio, United States